CLINICAL TRIAL: NCT06529484
Title: Investigation of the Effects of Foot Bath on Chemotherapy-Induced Fatigue in Pediatric Oncology Patients: A Randomized Controlled Trial
Brief Title: Foot Bath Effects on Chemotherapy-Induced Fatigue in Pediatric Oncology
Acronym: FBECIFPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Özge Eda Karadağ Aytemiz, Assistant Proffessor, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-22686390-050.99-46591
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nursing Caries
Keywords: Nursing, child, footbath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive interactive training and an educational booklet on fatigue, its definition, causes, development, coping strategies, and water temperature adjustment. Each patient gets a marked plastic basin for 8 liters and a thermometer.
  Starting the next day, patients will take a 38-40ºC warm water bath for 20 minutes between 21:00-22:00 nightly for 7 days to manage fatigue. This time ensures the child rests after the bath.
  In the initial 30-minute meeting, evaluation tools will assess the patient's personal and disease-related characteristics, fatigue level on the treatment day, impact due to fatigue, and coping strategies. Patients will be called daily for 7 days to assess fatigue levels using the Scale. On the 7th day, the final interview will use the 12-Item Scale and the Parental Fatigue Scale for 7-12 Year old patients.
  Interventions: Other: Warm Water Foot Bath Intervention
- Control Group (No Intervention): The control group will receive interactive training and an educational booklet covering the definition, causes, development, and effective coping strategies for chemotherapy-related fatigue. Patients in this group will be assessed between 21:00-22:00 in the evening, without the warm water foot bath intervention. The evaluations will focus on fatigue levels and other related outcomes over the 7-day period. On the 7th day, the final interview will use the 12-Item Pediatric Oncology Fatigue Scale and the Parental Fatigue Scale for 7-12 Year Old Pediatric Oncology Patients, concluding the study.

INTERVENTIONS:
Other: Warm Water Foot Bath Intervention — Participants will take a warm water foot bath at 38-40ºC for 20 minutes nightly for 7 days.
  Arms: Experimental Group

SUMMARY:
This study aims to evaluate the effects of foot baths on chemotherapy-induced fatigue in pediatric oncology patients. Current literature lacks studies assessing this intervention in the pediatric population. Chemotherapy, a common cancer treatment, often results in side effects such as nausea, vomiting, constipation, diarrhea, taste changes, mouth ulcers, and notably, fatigue. Fatigue affects 51-86% of pediatric cancer patients and significantly impacts their quality of life. Addressing fatigue comprehensively is crucial for improving patients' quality of life. Non-pharmacological methods like foot baths have shown promise in reducing chemotherapy-related fatigue. Previous studies with gynecological cancer patients and others have found that warm water foot baths can alleviate fatigue and improve relaxation by reducing sympathetic activity and facilitating oxygen and nutrient delivery to the brain. This randomized controlled trial is designed to scientifically evaluate the efficacy of foot baths in alleviating fatigue in pediatric patients post-chemotherapy.

DETAILED DESCRIPTION:
Study Objective: There are no existing studies in the literature that evaluate the effect of foot baths on chemotherapy-induced fatigue in the pediatric population. Therefore, this research aims to assess the impact of foot baths on fatigue in pediatric patients post-chemotherapy and scientifically examine this effect through a randomized controlled trial.

General Information: One of the commonly used treatment methods in coping with cancer is chemotherapy. Chemotherapy causes many side effects in patients, such as nausea and vomiting, constipation, diarrhea, changes in taste and smell, mouth ulcers, and notably, fatigue. Fatigue is frequently reported by patients. Literature indicates that 51-86% of children with cancer experience fatigue related to cancer and its treatment. Fatigue can negatively affect the quality of life of patients, making it an important area of focus in the care of children with cancer. Comprehensive management of fatigue is crucial for improving the patient's quality of life. One non-pharmacological method that can be used to reduce fatigue is a foot bath. In a study involving patients with gynecological cancer, soaking feet in warm water (41-42°C) for 20 minutes was found to be effective in reducing chemotherapy-related fatigue. Another study by Yamamoto and colleagues evaluating the physical and psychological effects of foot baths with warm water on cancer patients indicated that after a 5-minute massage with olive oil, soaking feet in water at 38-42°C for 20 minutes provided relaxation and pain relief by reducing sympathetic activity. Another study found that warm water foot baths facilitated the delivery of oxygen and nutrients to the brain by increasing blood volume through vasodilation, thus reducing fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Parents' consent to participate in the study and provide written informed consent.
* No diagnosed chronic illness other than cancer.
* Parents are literate in Turkish.
* Children aged between 7-12 years.
* Diagnosis of Stage 3 or 4 Non-Hodgkin Lymphoma.
* Receiving the first course of chemotherapy.
* Fatigue level of 3 or higher according to the Visual Fatigue Scale by the Oncology Nursing Society of America.

Exclusion Criteria:

* Children with cancer who have mental retardation and their parents.
* Children with cancer who have undergone surgical operations that hinder activities or result in significant organ loss, and their parents.
* Children with compromised skin integrity.
* Children with cancer and their parents who do not wish to participate in the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Parental Fatigue Scale Points | measured daily over a period of 7 days.
  The scale is designed to assess fatigue in pediatric oncology patients aged 7-12 years, as reported by their parents. It comprises 27 items and three subscales, with a total Cronbach's alpha value of 0.95, indicating high internal consistency. The subscales are as follows: General Problems: This subscale assesses general fatigue in pediatric oncology patients and includes items from the first and 18th questions. Sleep Problems: This subscale focuses on sleep-related issues stemming from fatigue, including items from the 19th to the 24th questions. Treatment-Related Problems: This subscale evaluates the impact of treatment on fatigue, covering items from the 25th to the 27th questions. The scale uses a Likert-type format, where responses are rated from "1" to "5," with "1" indicating "never" and "5" indicating "always." The total score ranges from a minimum of 27 to a maximum of 135 points. An increase in the scale score suggests a decrease in the child's level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Eda Karadağ Aytemiz, Principal Investigator — Koç University
Locations (1):
- Istanbul University-Cerrahpasa Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided